CLINICAL TRIAL: NCT07364019
Title: The Brain Health PRO Online Risk Factor Reduction Study for The Canadian Therapeutic Platform Trial for Multidomain Interventions to Prevent Dementia
Brief Title: The Brain Health PRO Online Risk Factor Reduction Study to Prevent Dementia
Acronym: BHPROOF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Alzheimer Society of Canada (Other); Baycrest (Other); The Canadian Consortium on Neurodegeneration in Aging (CCNA) (Unknown)
Responsible Party: Principal Investigator, Haakon Nygaard, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: H25-03523
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Dementia Prevention; Subjective Cognitive Impairment; Mild Cognitive Impairment; Cognitive Change; Lifestyle Intervention; Dementia Education
Keywords: dementia education; at risk for dementia; lifestyle intervention; dementia reduction; dementia risk factor; dementia prevention; cognitive impairment; Alzheimer risk
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This is a randomized delayed-start control trial examining the effects of the 6-month BHPro Intervention on modifiable lifestyle risk factors in older adults at risk for dementia. Participants will be randomized to either immediately receive the BHPro intervention or to the control group (6 month delayed start).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate BHPro Intervention Group (Experimental): Participants in this group will start Brain Health PRO immediately at baseline
  Interventions: Other: Brain Health PRO
- Delayed Start BHPro (Other): Participants in this group will start Brain Health PRO in 6 months (delayed)
  Interventions: Other: Brain Health PRO

INTERVENTIONS:
Other: Brain Health PRO — Immediate start of 6-month Brain Health PRO Intervention
  Other Names: BHPro
  Arms: Immediate BHPro Intervention Group
Other: Brain Health PRO — Delayed start of 6-month Brain Health PRO
  Other Names: BHPro
  Arms: Delayed Start BHPro

SUMMARY:
This study will recruit participants at risk for dementia to participate in an online educational program called Brain Health PRO (BHPro). The BHPro intervention is designed to address modifiable risk factors for dementia through a 6-month, fully online, educational program conveying the best available evidence for lifestyle changes that can mitigate dementia risk, and foster engagement toward one's own brain health. Achieving lifestyle changes in a diverse Canadian population through online education would be a major achievement in dementia prevention in Canada, with widespread personal and socioeconomic benefits.

Eligible participants will be randomly assigned to either start Brain Health PRO immediately or in 6 months (delayed-start control group). All participants will have the opportunity to have access to BHPro for 6 months during the course of the study and will have open access to all content for 12 months following the initial 6-month intervention. Participation will last from 18-24 months depending on group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Completion and documentation of the electronic Informed Consent Process (from the participant)
* Sufficient proficiency in English or French to undergo online assessments and participate in an online educational program.
* Technical ability to participate in an online educational program and remote assessments (i.e., regularly have access to a computer or tablet with an internet connection; have access to a desktop or laptop computer with an internet connection at least once every 6 months; ability to send and receive emails; ability to complete online assessments)
* Sufficient vision to participate in an online educational program and complete online cognitive testing
* Ages 50-80
* Classified as being at increased risk of dementia based on at least one of the following:

  * First-degree family history of dementia
  * Education level at or below high school (grade 12 or less)
  * Self-Reported: Hypertension, Hypercholesterolemia, Body Mass Index > 30 kg/m2 (derived from NIH Metric BMI Calculator), or Physical Inactivity (active is defined as engaging in a minimum of 20- 30 min of physical activity causing sweating and breathlessness, at least 2 times a week)

Exclusion Criteria:

* Individuals who have a clinical diagnosis of Dementia (based on self-report)
* Individuals who are currently participating in or have participated in a past study involving BHPro

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in modifiable risk factors as measured by a 7-item composite dementia risk factor score after 6 months. | Change from baseline to month 6
  The primary outcome is the change in a composite modifiable risk score comprised of the following 7 lifestyle risk questionnaires: Physical Activity, Nutrition, Sleep, Cognitive Engagement, Social and Psychological Health, Vascular Heatlh, and Vision and Hearing (each questionnaire is individually described under the secondary outcomes). Scores for each risk factor will be standardized (z-score transformation using cohort-wide mean and standard deviation at baseline). When necessary, scores will be multiplied by -1 so that positive scores reflect lower risk (e.g., greater engagement in physical activity). The participant-level mean risk score will be calculated which reflects the average z-score for the participant across the modifiable risk factors.

SECONDARY OUTCOMES:
Change in individual modifiable risk factors as measured separately by each of the 7 BHPro Lifestyle Risk Questionnaires after 6 months: Physical Activity | Change from baseline to month 6
  The International Physical Activity Questionnaire-Short Form is a brief 7-item self-report measure that captures types of and intensity of physical activity and sitting time. The total score is calculated by summing the accrued number of points assigned per question. The total score ranges between 0-9, with a higher score indicating more physical activity.
Change in individual modifiable risk factors as measured separately by each of the 7 BHPro Lifestyle Risk Questionnaires after 6 months: Nutrition | Change from baseline to month 6
  Shorter 11-item version of the Eating Pattern Self-Assessment Questionnaire developed by CCNA Team 5. The total score is calculated by calculating the accrued number of points assigned per question. The total score ranges between 0 and 22, with a higher score indicating more healthy eating habits.
Change in individual modifiable risk factors as measured separately by each of the 7 BHPro Lifestyle Risk Questionnaires after 6 months: Sleep | Change from baseline to month 6
  Brief 10-item questionnaire developed by BHPro sleep module content leads that assesses sleep duration, sleep patterns, and difficulties and daytime fatigue over the past 3 months. The total score is calculated by summing the accrued number of points assigned per question. The total score ranges between 1 and 20, with a higher score indicating healthier sleep.
Change in individual modifiable risk factors as measured separately by each of the 7 BHPro Lifestyle Risk Questionnaires after 6 months: Cognitive Engagement | Change from baseline to month 6
  A 6-item questionnaire assessing types and duration of cognitively engaging activities. The total score is calculated by summing the accrued number of points assigned per question. The total score ranges between 0 and 36, with a higher score indicating more cognitively stimulating activities.
Change in individual modifiable risk factors as measured separately by each of the 7 BHPro Lifestyle Risk Questionnaires after 6 months: Social and Psychological Health | Change from baseline to month 6
  An 8-item questionnaire comprising 1 item on loneliness, 1 item on ageism, 1 item on subjective age, 1 item on essentialist beliefs of aging and 4 items on depression, anxiety, stress, and social support from STOP-D. The total score is calculated by summing the accrued number of points assigned per question. The total score ranges between -1 and 50, with a higher score indicating poorer social and psychological health.
Change in individual modifiable risk factors as measured separately by each of the 7 BHPro Lifestyle Risk Questionnaires after 6 months: Vascular Health | Change from baseline to month 6
  12-item self-report questionnaire developed by the BHPro Vascular Health team based on the American Heart Association's Life's Simple Seven checklist of the main risk factors for heart disease and stroke. The total score is calculated by summing the accrued number of points assigned per question. The total score ranges between -4 and 8, with a higher score indicating better vascular health.
Change in individual modifiable risk factors as measured separately by each of the 7 BHPro Lifestyle Risk Questionnaires after 6 months: Vision and Hearing | Change from baseline to month 6
  10-item questionnaire developed by BHSP Vision and Hearing Module content leads that assesses perceived visual and auditory ability and actions taken to address potential vision/hearing difficulties. The total score is calculated by summing the accrued number of points assigned per question. If a user selects "Yes" for example, they receive 2 points for that question. The total score ranges between 0 and 20 points, with a higher score indicating poorer vision and hearing.
Change in self-efficacy as measured by the General Self-Efficacy Scale after 6 months. | Change from baseline to month 6
  Change in self-efficacy following participation in the study, as measured by the General Self-Efficacy Scale (GSE). The GSE measures perceived competence in dealing with a range of stressful or challenging situations. This self-report questionnaire contains 10-items, each rated on a 4-point scale (not true at all, hardly true, moderately true, exactly true). The total score is the sum of the scores for the 10 items, which is quantitative and ranges from 10-40, with a higher score indicating more self-efficacy.
Change in dementia literacy as measured by the Alzheimer's Disease Knowledge Scale after 6 months. | Change from baseline to month 6.
  Change in dementia literacy following participation in the study, as measured by the Alzheimer's Disease Knowledge Scale (ADKS). The ADKS is designed to assess knowledge about Alzheimer's Disease (AD) among laypeople, patients, caregivers, and professionals. This self-report questionnaire contains 30 true/false items. The total score is the sum of the scores from the 30 items, which is quantitative and ranges from 0-30, with a higher score indicating better knowledge about AD.
Change in cognition as measured by the Cogniciti Brain Health Assessment after 6 months. | Change from baseline to month 6
  The Cogniciti Brain Health Assessment (BHA) is a self-administered validated computerized cognitive assessment comprised of four tests (Spatial Working Memory, Stroop Interference, Face-Name Association, and Number-Letter Alternation). The overall Cogniciti Brain Health Assessment score ranges from 0-100 with a higher score indicating better cognition.

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Colubmia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes